CLINICAL TRIAL: NCT06262425
Title: Comparison of Different Repetitive Transcranial Magnetic Stimulation Protocols for Motor Learning in Healthy People. A Randomized Controlled Trial
Brief Title: rTMS Over S1 Enhance Motor Learning in Healthy People
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Neuron, Spain (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ALC001NR004
Record Dates: First submitted 2023-12-20; First posted 2024-02-16 (Actual); Last update posted 2025-09-02 (Actual); Status verified 2025-08

CONDITIONS: Transcranial Magnetic Stimulation; Motor Learning
Keywords: Transcranial magnetic stimulation; Motor learning; Somatosensory cortex; Motor function

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- repetitive Transcranial Magnetic Stimulation over primary somatosensory cortex (Experimental): Participants in the experimental group will receive 5 weekly sessions of repetitive Transcranial Magnetic Stimulation (rTMS) for two weeks. An excitatory stimulation over the primary somatosensory area corresponding to the dominant hand will be applied. For this purpose, the motor area will be localized and a coil will be placed 2 cm posterior to it. An isolated pulse will be applied to the motor area to ensure that the coil is not placed over the motor area using 110% of the motor resting threshold. After this, 22 trains of 10 Hz at an intensity of 90% of the motor resting threshold will be applied for 4 seconds, with a rest between series of 10 seconds (a total of 880 pulses). After the stimulation, participants will train with the Forced Response training program for a total of 500 correct repetitions and the Purdue Pegboard Test with 4 repetitions for right hand, left hand and both hands.
  Interventions: Device: repetitive Transcranial Magnetic Stimulation over primary somatosensory cortex
- repetitive Transcranial Magnetic Stimulation over primary motor cortex (Active Comparator): Participants in the active comparator group will receive 5 weekly sessions of repetitive Transcranial Magnetic Stimulation (rTMS) for two weeks. An excitatory stimulation over the primary motor cortex corresponding to the dominant hand will be applied. For this purpose, the motor area will be localized, and an isolated pulse will be applied to the motor area to ensure that the coil is placed over the motor area using 100% of the motor resting threshold. After this, 22 trains of 10 Hz at an intensity of 90% of the motor resting threshold will be applied for 4 seconds, with a rest between series of 10 seconds (a total of 880 pulses). After the stimulation, participants will train with the Forced Response training program for a total of 500 correct repetitions and the Purdue Pegboard Test with 4 repetitions for right hand, left hand and both hands.
  Interventions: Device: repetitive Transcranial Magnetic Stimulation over primary motor cortex
- Sham repetitive transcranial magnetic stimulation (Sham Comparator): Participants in the sham group will receive 5 weekly sessions of sham repetitive Transcranial Magnetic Stimulation (rTMS) for two weeks.To achieve the placebo, the localization of the area to be stimulated will be carried out but the coil will be placed in a vertical position so the current will not go through the skull and the patient will just feel the vibration, communicating to the participant that it is likely that during the stimulation process he/she will not feel anything. After the sham stimulation, participants will train with the Forced Response training program for a total of 500 correct repetitions and the Purdue Pegboard Test with 4 repetitions for right hand, left hand and both hands.
  Interventions: Device: sham repetitive Transcranial Magnetic Stimulation

INTERVENTIONS:
Device: repetitive Transcranial Magnetic Stimulation over primary somatosensory cortex — It will be applyed a magnetic field over the Somatosensory cortex of the patient that pretends to hiperexcite the membrans of the neurons inthis area to enhance motor learning
  Arms: repetitive Transcranial Magnetic Stimulation over primary somatosensory cortex
Device: repetitive Transcranial Magnetic Stimulation over primary motor cortex — It will be applyed a magnetic field over the primary motor cortex of the patient that pretends to hiperexcite the membrans of the neurons inthis area to enhance motor learning
  Arms: repetitive Transcranial Magnetic Stimulation over primary motor cortex
Device: sham repetitive Transcranial Magnetic Stimulation — It will be applied a sham stimulation with the same protocol that pretends to create the illusion of being stimulated
  Arms: Sham repetitive transcranial magnetic stimulation

SUMMARY:
The purpose of this study is to compare the effectiveness of different repetitive Transcranial Magnetic Stimulation protocols for enhancing motor learning in healthy peolple.

DETAILED DESCRIPTION:
This randomized clinical trial aims to compare the effectiveness of different repetitive Transcranial Magnetic Stimulation (rTMS) protocols in enhancing motor learning in healthy individuals. It focuses on two key brain areas: the primary motor cortex (M1) and the primary somatosensory cortex (S1), recognized for their roles in motor skill acquisition and execution.

Motor learning involves two distinct neural networks: the associative/premotor and sensorimotor networks. Studies suggest that the associative/premotor network predominates initially, followed by the sensorimotor network. M1 stores movement patterns, whereas S1 appears crucial for initial motor learning and movement adaptation.

rTMS, a non-invasive technique modulating neuronal excitability, has been used to improve motor function in patients with brain injuries. However, its effectiveness in healthy individuals has been variable, especially when stimulating M1 and S1. Prior research suggests that inhibitory rTMS in S1 may influence motor learning, but findings regarding its excitatory effect and comparison with M1 stimulation are mixed.

The primary hypothesis posits that excitatory rTMS in S1 will yield superior motor learning improvements compared to M1 stimulation in healthy individuals. The secondary hypothesis predicts improvements independent of the stimulated area.

The study will involve healthy participants, utilizing tests for accuracy and time. Methodology includes randomization, blind evaluation, and rTMS application based on assigned groups.

With a sample size of 35 subjects per group, data will be analyzed using parametric and non-parametric statistical tests to compare the effects of rTMS on M1 and S1 concerning motor learning in healthy subjects. Results will be considered significant with p < 0.05, and effect size will be evaluated.

This trial aims to provide clarity on the effectiveness of excitatory rTMS in specific brain areas to enhance motor learning in individuals without neurological pathologies, potentially impacting rehabilitation and motor performance.

ELIGIBILITY:
Inclusion Criteria:

* Older than 18 years old and younger than 65

Exclusion Criteria:

* Presenting any neurological pathology
* Pain during the study
* Any contraindications to rTMS, such as metal implants, history of epileptic seizures or taking medication that lowers the seizure threshold

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2024-01-20 (Actual); Primary Completion 2025-07-15 (Actual); Study Completion 2025-07-15 (Actual)

PRIMARY OUTCOMES:
Change in accuracy | Change from Baseline to 5 days and 10 days in accuracy
  Accuracy in associating one letter of the keyboard with a letter from the Phoenician alphabet presented in the screen. It will be measured by using the software PsychoPy, that has been used in other studies for measuring motor learning in an indirect way.

SECONDARY OUTCOMES:
Change in reaction time speed | Change from Baseline to 5 days and 10 days in reaction time speed
  Reaction time for responding correctly the association between one letter of the keyboard and a letter from the Phoenician alphabet presented in the screen. It will be measured by using the software PsychoPy, that has been used in other studies for measuring motor learning in an indirect way.
Change in pegs placed in 30 seconds | Change from Baseline to 5 days and 10 days in days placed in 30 seconds
  Number of pegs placed in a pegboard in 30 seconds will be measured. Patients will use just right hand first, after they will use just their left hand and finally with both hand at same time. This procedure will be repeated and average pegs placed in each condition will be noted. Purdue Pegboard Test will be used for measuring.

CONTACTS AND LOCATIONS:
Overall Officials: Alfredo Lerín Calvo, PhD student, Principal Investigator — Neuron, Spain
Locations (1):
- Neuron, Madrid, Madrid, Spain